CLINICAL TRIAL: NCT03373266
Title: Implication of Serum Fluoride Level Caused by Sevoflurane Versus Isoflurane Anesthesia Upon Renal Function After Kidney Transplantation.
Brief Title: Serun Fluoride and Kidney Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrady S Ibrahim, MD, Assistant professor, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB0000871242
Record Dates: First submitted 2017-12-02; First posted 2017-12-14 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Kidney Transplant; Complications
MeSH Terms: interventions — Sevoflurane; Isoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sevoflurane (Active Comparator): anesthesia was maintained with Sevoflurane 1-2%.
  Interventions: Drug: Sevoflurane
- isoflurane (Active Comparator): anesthesia was maintained with isoflurane 1-2%.
  Interventions: Drug: Isoflurane

INTERVENTIONS:
Drug: Sevoflurane — anesthesia was maintained with Sevoflurane 1-2%.
  Other Names: Inhalational anesthetic
  Arms: Sevoflurane
Drug: Isoflurane — anesthesia was maintained with isoflurane 1-2%.
  Other Names: Inhalational anesthetic
  Arms: isoflurane

SUMMARY:
Our primary goal is to investigate any hidden burden upon the grafted kidney from the increase of serum fluoride resulted from sevoflurane, versus isoflurane.

DETAILED DESCRIPTION:
Eighty patients with end stage renal failure undergoing living donor kidney transplant under general anesthesia were included in this study, by using an open (non-blinded) study design, patients were randomly assigned to two groups, 15 patients in each. Randomization was done through computer generated random tables. Isoflurane group; anesthesia was maintained with isoflurane 1-2%. Sevoflurane group; anesthesia was maintained with Sevoflurane 1-2%.

A peripheral intravenous access was secured in the hand opposite to the functioning fistula and induction of anesthesia was done with propofol 2mg/kg, neuromuscular blockade was maintained with atracurium 0.6mg/kg and all patients were intubated and ventilated to maintain end-tidal carbon dioxide (ETCO2) concentration between 30-40 mmHg. Anaesthesia was maintained with 1-2% isoflurane (isoflurane group) or 1-2% sevoflurane (sevoflurane group) with fresh gas flow of 2 L/min. In both groups inhalational anesthetic was delivered in an air-oxygen mixture of 1:1 ratio. Analgesia was maintained with fentanyl 1µg/kg/hr. Mannitol and sodium bicarbonate was given immediately before reperfusion (de-clamping of renal artery). Intraoperative monitoring included heart rate, noninvasive blood pressure, oxygen saturation, ETCO2, ECG and central venous line was placed in the right or left internal jugular vein depending upon the presence of dialysis catheter. Hemodynamic target include: mean arterial pressure of > 80mmHg, CVP between 10-15 mm Hg to optimize cardiac output and renal blood flow.

ELIGIBILITY:
Inclusion Criteria:

* end stage renal disease

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Serum fluoride | baseline before anesthesia
  Serum inorganic fluoride
Serum fluoride | one hour postoperative
  Serum inorganic fluoride
serum fluoride | 6 hours postoperative
  Serum inorganic fluoride
Serum fluoride | 12 hours postoperative
  Serum inorganic fluoride
Serum fluoride | 24 hours postoperative
  Serum inorganic fluoride
Serum fluoride | 48 hours postoperative
  Serum inorganic fluoride

SECONDARY OUTCOMES:
Serum creatinine | Baseline preoperative
  kidney function
Serum creatinine | 24 hours postoperative
  kidney function
Serum creatinine | 48 hours postoperative
  kidney function
Serum creatinine | one week postoperative
  kidney function
creatinine clearance | baseline before anesthesia
  kidney function
creatinine clearance | 24 hours postoperative
  kidney function
creatinine clearance | 48 hours postoperative
  kidney function
creatinine clearance | one week postoperative
  kidney function
Urine output | 24 hours postoperative
  kidney function
Urine output | 48hours postoperative
  kidney function

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrady S Ibrahim, M.D., Principal Investigator — assiut university faculty of medicine
Locations (1):
- Assiut university faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Burchardi H, Kaczmarczyk G. The effect of anaesthesia on renal function. Eur J Anaesthesiol. 1994 May;11(3):163-8. PMID 8050420